CLINICAL TRIAL: NCT07368660
Title: InPART Rx - Inpatient Provider Antibiotic Rate Benchmarking to Reduce Unnecessary Prescribing
Brief Title: InPART RX - Epicenters
Acronym: InPART RX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott K. Fridkin, Professor of Medicine and Epidemiology, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P009466; U54CK000601-01 (NIH); STUDY00003936 (Other: Emory IRB)
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hospital Infection; Standardized Antibiotic Prescribing Ratio (SAR)
Keywords: Stepped wedge; Stewardship; Hospitalists; Quality Metrics; Antibiotics Prescription; C. Difficile Infection (CDI)
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized approach of a quality improvement effort of peer comparative inpatient prescribing reports sent to hospitalists in 5 hospitals. The intervention will be rolled out sequentially to all 5 hospitals in 3-month intervals. The intervention will last 18 months at all 5 sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMS Providers (Experimental): Hospitalists will receive messages via email every 2 months with comparison data of the previous 2 months and antibiotic prescribing educational content.
  HMS providers will be receiving data on prescribing as part of the intervention.
  Interventions: Other: Messaging Hospitalists
- Usual Care Arm (Control) (Other): Hospitalists will receive bimonthly educational emails about simple steps to improve antibiotic prescribing.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Messaging Hospitalists — The intervention has two parts: (1) a one-time educational session on antibiotic de-escalation, and (2) bimonthly email feedback reports. Educational sessions, led by facility stewardship leads, focused on evidence-based recommendations for presumed pneumonia and urosepsis, specifically indications for empiric anti-pseudomonal coverage and use of Emory Healthcare's antibiotic prescribing assistance tool. Feedback reports reinforced these indications and provided a link to the tool.
  Arms: HMS Providers
Other: Usual Care — The usual care arm will be an educational email about simple steps to improve antibiotic prescribing sent bimonthly to all hospitalists.
  Arms: Usual Care Arm (Control)

SUMMARY:
InPART Rx is a collaborative research study to measure the impact of a planned quality improvement initiative to reduce unnecessary antibiotic prescribing by the Hospital Medicine Service through a process of receiving peer-comparison summary prescribing data bimonthly. The initiative is a collaboration between EHC Pharmacy, the School of Medicine (SOM) Division of Infectious Diseases, and the SOM Hospital Medicine Service.

Roughly one-third of antibiotics prescribed in the hospital setting are for the wrong dose, wrong drug, or wrong duration, resulting in considerable unnecessary antibiotic exposure among the inpatient population. Such use increases patient risk for adverse events such as infectious diarrhea or antibiotic-resistant infections. Inpatients cared for by Hospital Medicine providers are a growing proportion of all patients, and developing efficient techniques to reduce unnecessary antibiotic prescribing by these providers would benefit this growing population of patients.

The research team aims to measure the impact of implementing a process to provide peer comparisons of antibiotic prescribing among Hospitalists at four Emory Healthcare (EHC) hospitals back to these providers in an effort to minimize unnecessary antibiotic prescribing. All 147 current Hospital Medicine Service providers will participate as part of the Division's quality improvement effort, receiving no compensation. Only summary patient encounter information without private health insurance (PHI) will be presented back to the providers; investigators will track changes in summary prescribing metrics and summary patient outcomes every month. If such an automated peer-comparison feedback process is effective in safely reducing unnecessary antibiotic prescriptions in EHC, similar processes may be adapted to other inpatient provider groups or serve as a model for other healthcare systems.

The goal of this quality improvement (QI) work is to use traditional QI methods of peer-comparison through data feedback to improve antibiotic prescribing among EHC HMS by reducing unnecessary antibiotic use and improving patient safety on the EHC HMS.

DETAILED DESCRIPTION:
The intervention is messaging to hospitalists via email every 2 months (bi-monthly) that contains peer comparison data of the previous 2 months and antibiotic prescribing educational content.

The details of the content may include a relative rank in prescribing metrics, with blinding to specific peers' identities, and department-wide and facility-specific goals highlighted. Those in the lowest prescribing quartile will earn the designation of "Top Performer". The usual care arm will be an educational email about simple steps to improve antibiotic prescribing sent bimonthly to all hospitalists.

Data Sources: The primary source of data will be the Emory Hospital (EH) Clinical Data Warehouse (CDW), a repository that integrates data from multiple clinical applications within EHC and has the flexibility to create customized, research-specific metrics for all adults (≥18 years old) admitted to the HMS at either Emory University Hospital (EUH), Emory University Hospital Midtown (EUHM), Emory Johns Creek Hospital (EJCH), or Emory St. Joseph's Hospital (ESJH).

ELIGIBILITY:
Inclusion Criteria:

* All Hospital Medicine Service (HMS) Providers at either Emory University Hospital (EUH), Emory University Hospital Midtown (EUHM), Emory Johns Creek Hospital (EJCH), or Emory St. Joseph's Hospital (ESJH)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Observed provider-specific antibiotic prescribing rate | Baseline and bimonthly for 2 years
  The observed provider-specific antibiotic prescribing rate is defined as the billed days of therapy (DOT) of Broad-Spectrum, Hospital-Onset (BS-HO) antibiotics per 1000 billed patient-days.

SECONDARY OUTCOMES:
C. difficile infection | Up to 8 weeks post discharge (9 weeks from admission on average)
  C. difficile infection occurring during inpatient stay (average 7 days) or within 8 weeks after discharge among patients managed by hospital medicine and discharged with an ICD-10 diagnosis code for community-acquired pneumonia, urinary tract infection (UTI), or urosepsis.
Number of participants with a prolonged length of initial hospital stay | Hospital stay, an average of 10 days
  Prolonged initial hospital stays, defined as a length of stay exceeding 7 days from arrival at the emergency department (ED) to hospital discharge, among patients managed by hospital medicine and discharged with an International Classification of Diseases (ICD)-10 diagnosis code for community-acquired pneumonia, urinary tract infection (UTI), or urosepsis.
In-hospital mortality | Hospital admission, an average of 7 days
  Rate of in-hospital mortality among patients managed by hospital medicine and discharged with an ICD-10 diagnosis code for community-acquired pneumonia, urinary tract infection (UTI), or urosepsis.
Hospital readmissions | 30 days after hospital discharge
  Hospital readmissions up to 30 days after index hospital discharge among patients managed by hospital medicine and discharged with an ICD-10 diagnosis code for community-acquired pneumonia, urinary tract infection (UTI), or urosepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K. Fridkin, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown (EUHM), Atlanta, Georgia
  - Emory University Hospital (EUH), Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: No